CLINICAL TRIAL: NCT06749509
Title: Effects of Musculoskeletal Rehabilitation Courses on Work Ability (Tules-kurssit Ja Työkyky)
Brief Title: Effects of Musculoskeletal Rehabilitation Courses on Work Ability
Status: Enrolling by invitation | Type: Observational
Sponsor: Social Insurance Institution, Finland (Other)
Collaborators: Finnish Institute of Occupational Health (Other)
Responsible Party: Sponsor
Other Study IDs: KELA_4822_2024
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Diseases or Conditions; Musculoskeletal Disorders
Keywords: Musculoskeletal Diseases; Musculoskeletal Disorders; Work Ability; Rehabilitation; Telerehabilitation; Quality of Life; Pain; Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Pain; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Face-to-face musculoskeletal rehabilitation (A): Participation in a face-to-face rehabilitation course organized by the Social Insurance Institution of Finland (Kela) for those with musculoskeletal disorders (MSD) (A)
  Interventions: Other: Face-to-face musculoskeletal rehabilitation
- Musculoskeletal telerehabilitation (B): Participation in a telerehabilitation course organized by Kela for those with MSD (B)
  Interventions: Other: Musculoskeletal telerehabilitation
- Controls (C): Persons with MSD who had contacted their occupational health care because of musculoskeletal symptoms, and will not participate in Kela's musculoskeletal rehabilitation course during the study period
  Interventions: Other: Controls

INTERVENTIONS:
Other: Face-to-face musculoskeletal rehabilitation — Kela's rehabilitation course for those with MSD includes two 5-day periods and one 3-day period of face-to-face rehabilitation, which are carried out in a Finnish rehabilitation center over a 9-month period and implemented by a multidisciplinary team of rehabilitation experts. The rehabilitation course is group-based and provided free of charge. The 9-month rehabilitation period also includes calls to the participants before and after rehabilitation. The course is intended for persons over the age of 18 with diagnosed MSD and difficulties coping with work or studies. The course provides support, tools, and coaching to help manage daily life and work with MSD. Self-rehabilitation is an important component of the program. Individual goals based on the GAS method are set, evaluated, and adjusted during the rehabilitation. A medical statement is required when applying for the rehabilitation course.
  Groups: Face-to-face musculoskeletal rehabilitation (A)
Other: Musculoskeletal telerehabilitation — Kela´s MSD telerehabilitation course is arranged entirely as telerehabilitation, and it includes videoconferencing, online rehabilitation, and group-based rehabilitation days implemented by a multidisciplinary team of rehabilitation experts. Participation does not require particular IT skills, but appropriate equipment (e.g., mobile phone, laptop, tablet computer) is needed. The rehabilitation course is free of charge, and the total duration, including the calls before and after rehabilitation, is approximately 7 months. The course is intended for persons over the age of 18 with diagnosed MSD and difficulties coping with work or studies. The course provides support, tools, and coaching to help manage daily life and work with MSD. Self-rehabilitation is an important component of the program. Individual goals based on the GAS method are set, evaluated, and adjusted during the rehabilitation. A physiotherapist's recommendation is required when applying for the telerehabilitation course
  Groups: Musculoskeletal telerehabilitation (B)
Other: Controls — The control participants have an MSD diagnosis and musculoskeletal symptoms. Based on an occupational physiotherapist's brief evaluation they are eligible to apply for Kela's musculoskeletal rehabilitation (the interventions below). By them own choice, however, they will not participate in these rehabilitation programs in the near future. The controls are recruited via two occupational health care producers in the private sector.
  Groups: Controls (C)

SUMMARY:
The goal of this observational study is to learn about the effects of two different musculoskeletal rehabilitation programs in working-age people with musculoskeletal disorders. The main question it aims to answer is:

Do musculoskeletal rehabilitation programs A or B improve work ability in people with musculoskeletal disorders?

Participants starting in rehabilitation programs A and B will answer survey questions about their work ability and related factors three times: when starting, immediately after the rehabilitation ends, and 4 months after ending the rehabilitation. Participants in study group C will answer the same questions during the same time period.

Researchers will compare participants in rehabilitation programs A and B to participants in group C, who have musculoskeletal disorders but will not participate in rehabilitation programs. The comparison is done to see if there are differences in the changes in work ability and related factors, such as pain or quality of life.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 ja 2:

* diagnosed musculoskeletal disorder
* 18 years or older
* in employment, returning to work, studying, or receives rehabilitation subsidy
* participating in either of the following:

  * Kela's face-to-face musculoskeletal rehabilitation (A)
  * Kela's musculoskeletal telerehabilitation (B)
* willingness to participate in the study

Group 3 (Controls):

* diagnosed musculoskeletal disorder
* 18 years or older
* in employment, returning to work, studying, or receives rehabilitation subsidy
* musculoskeletal symptoms have lasted at least 3 months and the person has participated in physiotherapy or self-rehabilitation without satisfactory results
* willingness to participate in the study

Exclusion Criteria:

Group 3 (Controls):

* Current rehabilitation needs are related to post-treatment care or post-discharge rehabilitation.
* acute or untreated substance use disorder
* participating in or apply for Kela's musculoskeletal rehabilitation services (A or B) during the next few months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those starting in either of the following services between January 2025 and January 2026:
  * Kela's face-to-face musculoskeletal rehabilitation (A)
  * Kela's musculoskeletal telerehabilitation (B).
  Persons with MSD who contacted their occupational health care between January 2025 and January 2026 because of musculoskeletal symptoms, but will not participate in Kela's musculoskeletal rehabilitation. Two private companies offering occupational health care services nationally are involved.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Work Ability at 4-6 Months and 8-10 Months | Baseline (pre-intervention), 4-6 months (after the intervention), 8-10 months (4-month follow-up)
  Work Ability Index questionnaire (7-49 points; the higher score indicates better work ability)

SECONDARY OUTCOMES:
Change from Baseline in Mood at 4-6 months | Baseline (pre-intervention), 4-6 months (after the intervention)
  Beck's Depression Inventory (BDI-21) (0-63; the higher score indicates more depressive symptoms)
Change from Baseline in Quality of Life at 4-6 months | Baseline (pre-intervention), 4-6 months (after the intervention)
  World Health Organization Quality of Life Instrument (WHOQOL-BREF) (0-100; the higher score indicates better quality of life)
Change from Baseline in Functional Ability at 4-6 months | Baseline (pre-intervention), 4-6 months (after the intervention)
  PROMIS®-29 Profile v2.1 (without 4 questions concerning depression) (t-score; the higher score indicates more measured quality)
Change from Baseline in Pain at 4-6 months and 8-10 months | Baseline (pre-intervention), 4-6 months (after the intervention), 8-10 months (4-month follow-up)
  5 questions from PROMIS®-29 Profile v2.1 concerning pain and 5 questions concerning musculoskeletal pain characteristics
Change from Baseline in Return-to-Work Self Efficacy at 4-6 months | Baseline (pre-intervention), 4-6 months (after the intervention)
  Return-to-Work Self Efficacy (RTW-SE), modified version (0-66; the higher score indicates better self efficacy)
Invidual Goal Achievement | 4-6 months (after intervention)
  Goal Attainment Scaling method (GAS)
Days Lost Through Sickness | Between January 1, 2024 and June 30, 2026
  Register-based data concerning sickness allowance. The sickness allowance is paid as compensation for loss of income due to incapacity for work lasting less than a full year. Periods which have lasted ten days or more are available in Kela's register.

CONTACTS AND LOCATIONS:
Locations (1):
- The Social Insurance Institution of Finland, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No